CLINICAL TRIAL: NCT06088758
Title: Normothermic Machine Perfusion of Steatotic Livers for Expansion of Donor Organ Pool
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Heidi Yeh, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023P002561
Record Dates: First submitted 2023-09-22; First posted 2023-10-18 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Liver Transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Liver Transplantation with Steatotic Liver (Experimental): Graft will be selected if 30-60% macrosteatosis and transplanted into liver transplant recipient with MELD of 15-25.
  Interventions: Device: Normothermic machine perfusion (NMP) of steatotic liver

INTERVENTIONS:
Device: Normothermic machine perfusion (NMP) of steatotic liver — Steatotic liver grafts that are selected will be run on NMP to assess quality of graft and determine whether it meets criteria for transplantation

SUMMARY:
The goal of this clinical trial is to assess the ability of Normothermic Machine Perfusion (NMP) to resuscitate moderately steatotic livers for transplantation in patients. This will be a single-site clinical trial placing donor livers with 30-60% macrosteatosis on NMP, and then transplanting those that meet commonly accepted viability criteria. The results of this study could lead to a trial extending NMP transplantation to severely steatotic livers, further expanding the donor organ pool.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Listed for liver transplantation at MGH
* Calculated MELD-Na score <= 25
* Able to consent

Exclusion Criteria:

* Status 1a
* Cardiac or pulmonary disease
* Prior liver transplant
* Requiring pressors at the time of liver offer
* MELD<15 and asymptomatic from liver disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Early allograft dysfunction | First week after transplant
  Number of participants with initial poor function of liver allograft: measured by presence of 1 or more of the following: aspartate aminotransferase (AST) level higher than 2000 IU/L (to convert to microkatals per liter, multiply by 0.0167) within the first 7 postoperative days; bilirubin 10 mg/dL or higher (to convert to micromoles per liter, multiply by 17.104) on postoperative day 7; international normalized ratio (INR) of 1.6 or higher on postoperative day 7; or graft primary nonfunction within the first 7 days, defined as irreversible graft dysfunction leading to recipient death or emergency retransplant, in the absence of immunologic or surgical causes

SECONDARY OUTCOMES:
Intraoperative inotropic support | At reperfusion, 15 minutes, 1 hour, 2 hours, and 3 hours after reperfusion
  Number of participants in need of inotropic support to maintain hemodynamics intraoperatively after reperfusion of liver allograft
Need for post-operative inotropic support | First 30 days post-transplantation
  Number of participants in need of inotropic support upon admission to the ICU
Length of post-operative inotropic support | First 30 days post-transplantation
  Length of inotropic support used after admission to the ICU, if needed
Need for post-operative mechanical ventilation | First 30 days post-transplantation
  Number of participants in need of mechanical ventilation upon admission to ICU
Length of post-operative mechanical ventilation | First 30 days post-transplantation
  Length of intubation after admission to ICU, if mechanical ventilation needed
ICU length of stay | First 30 days post-transplantation
  Length of stay in ICU post-transplant
Renal replacement therapy requirement | First 30 days post-transplantation
  Number of participants who require renal replacement therapy during the first 10 days after liver transplantation, if not on renal replacement prior to transplant
Peak AST and ALT | First 7 days post-transplantation
  Concentration of peak AST and ALT
Internal Normalized Ratio (INR) | First 7 days post-transplantation or within first 30 days post-op if discharge is longer than 7 days out
  INR measurements for each participant until post-op day 7 or discharge
Total bilirubin | First 7 days post-transplantation or within first 30 days post-op if discharge is longer than 7 days out
  Total bilirubin measurement (mg/dl) on post-op day 7 or day of discharge
30-day patient survival | First 30 days post-transplantation
  30-day patient survival (percentage)
Re-listing for transplantation | First 30 days post-transplantation
  Number of participants who require re-listing for liver transplantation within 30 days post-op
Adverse events | First 30 days post-transplantation
  Incidence of any additional adverse events, not including 24-hour ICU stay post-transplant, post-transplant transfusion <=6 units pRBCs, <=2 units FFP, <=2 units 6-pack of platelets, as these are considered routine
Biopsy-proven rejection episodes | Assessed at 3, 6, and 12 months post-transplant
  Number of participants with biopsy-proven rejection episodes
Liver function tests more than 3 times normal | Assessed at 3, 6, and 12 months post-transplant
  Number of participants with liver function tests more than 3 times normal; liver function tests (LFTs) will measure AST/ALT, bilirubin, INR
Additional procedures | Assessed at 3, 6, and 12 months post-transplant
  Number of participants that require additional procedures beyond normal recovery standard of care post-liver transplant
Re-admissions | Assessed at 3, 6, and 12 months post-transplant
  Number of participants with re-admissions after initial discharge
Ischemic cholangiopathy and anastomotic strictures by imaging | Assessed at 3, 6, and 12 months post-transplant
  Number of participants with evidence of ischemic cholangiopathy and anastomotic strictures by imaging
Vascular complications by cross-sectional imaging or angiography | Assessed at 3, 6, and 12 months post-transplant
  Number of participants with evidence of vascular complications by cross-sectional imaging or angiography
Presence of steatosis by imaging or histology | Assessed at 3, 6, and 12 months post-transplant
  Number of participants with evidence of steatosis by imaging or histology
Degree of steatosis by imaging or histology | Assessed at 3, 6, and 12 months post-transplant
  Degree of steatosis by imaging or histology, if present
Renal dysfunction | Assessed at 3, 6, and 12 months post-transplant
  Presence of a decrease in GFR > 40 from pre-transplant baseline or creatinine >2 if received simultaneous liver-kidney transplant
Hyperlipidemia | Assessed at 3, 6, and 12 months post-transplant
  Number of participants with evidence of hyperlipidemia
Immunosuppression medications | Assessed at 3, 6, and 12 months post-transplant
  Types of immunosuppression medications required
Dosage of immunosuppression medications | Assessed at 3, 6, and 12 months post-transplant
  Dosage of immunosuppression medications required in respective unit measurement (i.e. milligrams)
Drug levels of immunosuppression medications | Assessed at 3, 6, and 12 months post-transplant
  Drug levels of immunosuppression medications present in blood titers drawn from participant in respective unit measurement (i.e. ng/mL)
Re-listing for transplantation | Assessed at 3, 6, and 12 months post-transplant
  Number of participants who require re-listing for transplantation within 1 year post-op
Graft failure | Assessed at 3, 6, and 12 months post-transplant
  Number of participants with evidence of graft failure
Patient death | Assessed at 3, 6, and 12 months post-transplant
  Number of participants with evidence of patient death

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Brigham, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No